CLINICAL TRIAL: NCT01754909
Title: Mitigation of Radiation Pneumonitis and Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CLIN-004-12S; 1I01CX000569-01A2 (NIH)
Record Dates: First submitted 2012-11-29; First posted 2012-12-21 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Lung Cancer; Radiation Pneumonitis
Keywords: lung cancer; radiation pneumonitis; mitigation; enalapril; placebo
MeSH Terms: conditions — Lung Neoplasms; Radiation Pneumonitis | interventions — Enalapril

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- enalapril (Active Comparator): Use of enalapril in subjects undergoing radiotherapy for lung cancer.
  Interventions: Drug: Enalapril
- placebo (Placebo Comparator): Use of placebo in subjects undergoing radiotherapy for lung cancer
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Enalapril — Enalapril once a day, orally, as 2.5 , 5, or 10 mg tablets to be given in escalating doses, to subjects undergoing radiotherapy for lung cancer
  Arms: enalapril
Drug: placebo — Placebo, once a day, orally, as 2.5 , 5, or 10 mg tablets to be given in escalating doses, to subjects undergoing radiotherapy for lung cancer
  Arms: placebo

SUMMARY:
This project will test the effect of enalapril to mitigate the lung damage that can occur as a side effect of radiation therapy for lung cancer or other intrathoracic cancers. Thousands of Veterans develop lung cancer every year, and are treated by radiation therapy. Studies of lung radiation injury in laboratory animals show that with enalapril, investigators can significantly reduce the severity of radiation injury to the lung. Enalapril is FDA approved and in common use for treatment of hypertension, kidney disease, and heart failure. These studies will advance that work to human use. Successful mitigation of lung radiation damage will improve the quality of life in Veterans and non-Veterans who are treated for lung cancer by radiation, and may also improve cure rates of radiation therapy for lung cancer.

DETAILED DESCRIPTION:
Aim 1: To test the benefit of enalapril, an angiotensin-converting-enzyme-inhibitor, to mitigate radiation pneumonitis and fibrosis in humans.

Subjects

Men and women undergoing radiation therapy for lung cancer or other intrathoracic cancers at the Baltimore the Milwaukee or Ann Arbor Veterans Affairs Hospital are eligible. Subjects will be recruited to this phase 2 trial after their diagnosis of cancer and after referral to Radiation Oncology for treatment. The existence of this study will be posted in the Radiation Oncology clinics. Dr Cohen, Dr Beth Gore, and Dr Michelle Mierzwa (co-investigators) and our study coordinators will ensure recruitment. The informed consent process will be done by Dr Cohen or Gore or Dr Mierzwa or the study coordinators. Subjects who require radiation therapy to attempt to cure or to palliate their disease will be eligible for this study. Subjects eligible for surgical resection and who do not need radiation therapy will not be eligible for this study. Subjects on ACE inhibitors, angiotensin blockers, or renin antagonists will be excluded. Use of other antihypertensives is not an exclusion criterion. There will be no inclusion or exclusion by race or ethnic origin. Women and minorities are eligible. Children are not eligible because children do not develop lung cancer. Previous surgery and past or current use of chemotherapy are not exclusions. Subjects will have a Karnofsky performance status >/=70, absolute neutrophils > 1000/mm^3, platelets > 75,000/mm^3, and hematocrit > 25%. Liver and kidney function tests will be within normal range and baseline blood pressure will be systolic > 110 mmHg sitting. Pregnant or nursing subjects are excluded and fertile patients will use contraception. Lung function tests including spirometry, lung volumes and diffusing capacity will be obtained as part of standard of care for patients prior to radiotherapy, but indices from lung function tests will not be a cause for exclusion.

The mean lung dose will be >/= 18 Gy and/or V20 >20%. Radiation will be delivered with standard fractionation schedule of 1.8 to 2 Gy per day, 5 days per week, without planned treatment breaks.

Experimental design

Radiation treatment starts at time 0, and is given to completion, as indicated. Enalapril or placebo are started after the first radiation treatment fraction and continued thereafter. The renin-angiotensin system is tested at time 0, at three weeks, and at the completion of radiation treatment. CT scanning is done at time 0 and every three months thereafter for the first two years. Median survival is expected to be 18 months.

Subjects will undergo therapeutic irradiation as indicated for clinical care. They will be enrolled to this masked, phase 2 trial at the start of radiation therapy (RT), stratified for cancer stage, then randomized to enalapril or identical-appearing placebo. Randomization will be done by the Department of Biostatistics, Medical College of Wisconsin, using random number tables; the center pharmacies will be notified of the assignment to enalapril or placebo. There will be no stratification by age, gender, lung cancer histology, or use of chemotherapy since these do not have a consistent relation with the occurrence of RP . Use of enalapril or placebo will not be known to the patients or their physicians during the time of study. The medical center pharmacy will stock and provide the study drug. Study drug, enalapril or placebo, will be started after the first fraction of the RT, at 2.5 mg by mouth once a day and increased to 10 mg/day in weekly increments as tolerated. Routine clinical care during the course of irradiation includes weekly or more frequent clinical assessment and vital signs. Blood testing for kidney function and potassium will occur within ten days after start of study drug. Additional patient visits will not occur for this study alone. Additional blood testing will occur in usual clinical care and will also be recorded. Routine care, independent of this study, includes CT scan chest imaging every three months for the first two years of follow-up. The study drug will be continued for life.

Endpoints for injury

The primary endpoint is symptomatic grade 2 or higher radiation pneumonitis, as defined by the established criteria, within the first 4 months of irradiation. The NCI Common Terminology Criteria Adverse Event (CTCAE) version 4.0 will be used to grade pulmonary toxicity. CTCAE is a worldwide standard for reporting adverse events from all modalities on cancer clinical trials. Pneumonitis is a new-onset and persistent cough requiring anti-tussive agents and or dyspnea with effort that is unexplained by other pulmonary illness. It may last for days to weeks. Severe cases may evolve to respiratory failure. Use of such patient-reported symptoms is strongly recommended for cancer-related clinical trials. Radiographic changes of RP occur in over half of subjects undergoing therapeutic thoracic irradiation; radiographic RP will be a secondary endpoint. Classic radiographic manifestations of RP are increased lung density within the radiation field within the first six months after radiation therapy that is not explained by infection or cancer. radiographic pneumonitis will be recorded by two investigators (Drs Gore and Antonescu-Turcu, EG, AAT), using the scale reported by Guckenberger. Investigators expect a radiographic rate of RP of 50%.

Investigators expect almost all surviving subjects to have fibrosis by CT scanning at 6 and 12 months, and will test this as another major endpoint. Radiation fibrosis in the lung is evident as scarring with volume loss and bronchiectasis within the radiation field at six months or more after radiation therapy, not explained by infection or cancer. radiographic fibrosis will be recorded and quantified by two investigators (EG, AAT). Reduction in diffusion capacity for carbon monoxide (DLCO) correlates with pulmonary radiation fibrosis. DLCO is obtained in all survivors at the 12 month time point, and will be compared to baseline values as an additional secondary endpoint. The occurrence of clinical grade 2 or higher RP, of radiographic RP and fibrosis as dichotomous variables, will be compared for the subjects on enalapril compared to those on placebo. For RP, any image showing RP will assign a subject to the RP group. For fibrosis, the last CT scan will be used.

Investigators will test quality of life as a secondary endpoint. The Functional Assessment of Cancer Therapy -lung (FACT-L version 4) will be used to assess Quality of Life (QoL). FACT-L contains four general (physical, social/family, emotional, and functional well being) and one lung cancer specific subscale. QoL will be assessed pretreatment, and at 12 months post treatment. Use of patient-reported data is strongly recommended for cancer-related clinical trials.

Aim 2: To test the mechanism of mitigation by enalapril

Subjects These are the same subjects as in aim 1.

Experimental design Investigators will test the major components of the renin-angiotensin system; angiotensinogen, plasma renin activity, and angiotensin II (ang II). These will be measured at baseline, at three weeks after the start of irradiation, and at the completion of irradiation. Investigators will test their mechanistic involvement by their change with use of enalapril, in particular whether the benefit of enalapril is correlated with its effect to lower the plasma ang II levels. Other components of the RAS, including angiotensin (1-7), aldosterone, AcSDKP, and bradykinin will not be tested because experimental studies have not shown them to be relevant to mitigation of normal tissue radiation injury.

Baseline elevation of one or more of these RAS components, compared to known levels in the normal population, may correlate with development of RP and or fibrosis in the control, placebo group. This may permit better focused use of mitigators in the future, in only those at risk.

Enalapril, by inhibition of ACE, will reduce plasma ang II and lead to a feedback elevation of PRA. This will confirm adherence to drug therapy and may also correlate with its benefit. Elevation of PRA in subjects on enalapril, but without mitigation benefit, will show that it is ineffective, despite its adequate bioavailability.

Aim 3: To confirm that enalapril does not adversely affect cancer treatment outcomes.

Subjects These are the same subjects as in aim 1.

Experimental design Investigators will compare cancer recurrence and cancer-related survival in subjects on enalapril versus placebo. Cancer recurrence will be assessed clinically, as confirmed by CT imaging and or histology. The RECIST criteria will be used. Recurrence rates and survival will be assessed by interim safety analyses during the study, and finally at its completion. In the statistical analysis, investigators will account for the effects of interim sampling for the safety analyses, and will adjust for patient and disease characteristics as well as missing data. A benefit of enalapril on RP may enhance patient survival. An adverse effect of enalapril on survival will stop this study. But a cohort of 162 Veterans showed no difference in patient survival for those on ACE inhibitor compared to those not on ACE inhibitor. Thus, investigators do not expect adverse changes in recurrence rates or patient survival.

Expected results, potential problems, and long-term impact

Investigators expect that subjects on enalapril will have significantly less clinical and radiographic RP and fibrosis, compared to those on placebo. Investigators expect that subjects on placebo who develop RP and or fibrosis may have baseline elevation of AGT and PRA compared to those who don't develop RP and or fibrosis, and that the mitigation benefit of enalapril will correlate with its effect to increase the PRA and reduce the plasma ang II levels. Investigators expect that enalapril will not increase cancer-related mortality, and may even enhance overall patient survival through mitigation of radiation lung injury.

ELIGIBILITY:
Inclusion Criteria:

* Men and women undergoing radiation therapy to the chest for cancer at the Baltimore, the Milwaukee, and Ann Arbor Veterans Affairs Hospital are eligible.
* Subjects who require radiation therapy to attempt to cure or to palliate their disease will be eligible for this study.

Exclusion Criteria:

* Subjects eligible for surgical resection and who do not need radiation therapy will not be eligible for this study.
* Subjects who must remain on ACE inhibitors, angiotensin blockers, or renin antagonists will be excluded.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric P Cohen, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (3):
- United States (3):
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kharofa J, Cohen EP, Tomic R, Xiang Q, Gore E. Decreased risk of radiation pneumonitis with incidental concurrent use of angiotensin-converting enzyme inhibitors and thoracic radiation therapy. Int J Radiat Oncol Biol Phys. 2012 Sep 1;84(1):238-43. doi: 10.1016/j.ijrobp.2011.11.013. Epub 2012 Jan 31. PMID 22300564
- [Result] Citrin DE, Prasanna PGS, Walker AJ, Freeman ML, Eke I, Barcellos-Hoff MH, Arankalayil MJ, Cohen EP, Wilkins RC, Ahmed MM, Anscher MS, Movsas B, Buchsbaum JC, Mendonca MS, Wynn TA, Coleman CN. Radiation-Induced Fibrosis: Mechanisms and Opportunities to Mitigate. Report of an NCI Workshop, September 19, 2016. Radiat Res. 2017 Jul;188(1):1-20. doi: 10.1667/RR14784.1. Epub 2017 May 10. PMID 28489488

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 consented
Pre-assignment Details: Verification of eligibility.
  Seven did not start study drug. Six of those because found ineligible after enrollment. One of those because of early termination of study.
Period: Overall Study
Arm/Group | Enalapril | Placebo
Started | 20 | 23
Completed | 20 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enalapril | Placebo | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 10 | 13 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 20 | 22 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 23 | 43
absence of pneumonitis or fibrosis [Count of Participants; unit: Participants] — as per clinical asessment
  Participants | 20 | 23 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Radiation Pneumonitis
Description: The clinical occurrence and grade of radiation pneumonitis, by National Cancer Institute Common Terminology Criteria Adverse Event grading ( NCI CTCAE)
Time Frame: two years
Measure: Number; unit: participants
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 20 | 23
participants | 8 | 10
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority — Occurrence rates, comparison by t test; p = 0.05, t-test, 2 sided

2. Secondary Outcome: Number of Participants With Radiation Pneumonitis by CT Scan
Description: The occurrence and grade of radiation pneumonitis by radiographic criteria, using CT scanning
Time Frame: six months
Population: analyzed by CT scan readings done in a masked fashion
Measure: Count of Participants; unit: Participants
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 20 | 21
Participants | 16 | 12

3. Secondary Outcome: Number of Participants With Radiation Fibrosis
Description: The occurrence and grade of radiation fibrosis by radiographic criteria, using CT scanning
Time Frame: one year
Measure: Number; unit: participants
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 20 | 23
participants | 8 | 4

ADVERSE EVENTS:
Time Frame: lifetime of subject or until study end April 2018, an average of 2 years
Description: Hospitalization or death
Arm/Group | Enalapril | Placebo
All-Cause Mortality (participants affected / at risk) | 11/20 | 7/23
Serious Adverse Events (participants affected / at risk) | 9/20 | 11/23
Other Adverse Events (participants affected / at risk) | 7/20 | 8/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enalapril (N=20) | Placebo (N=23)
death or hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 11 (11)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enalapril (N=20) | Placebo (N=23)
hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 8 — not death

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT01754909/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT01754909/SAP_001.pdf